CLINICAL TRIAL: NCT02690064
Title: Mechanisms for Vascular Dysfunction and Exercise Tolerance in CF
Acronym: CF-AOX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Ryan Harris, Principal Investigator, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CF-AOX
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cystic Fibrosis
Keywords: Endothelial Function; Maximal Exercise Capacity; Flow Mediated Dilation; Antioxidant; FEV1
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ascorbic Acid; Vitamin E; Thioctic Acid; Resveratrol; mitoquinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acute Antioxidant Treatment (Experimental): Following an overnight fast, blood samples, flow-mediated dilation, lung function, and exercise capacity (VO2 peak) (post only) will be performed at baseline and 2 hours following either a single dose oral 1) antioxidant cocktail (1000 mg Vitamin C, 600 IU vitamin E, 600 mg Alpha Lipoic Acid) 2) Resveratrol (1500 mg) 3) Mitoquinol (10 mg) or placebo on two days separated by at least 72 hours.
  Interventions: Dietary Supplement: Acute Antioxidant; Other: Placebo
- Chronic Antioxidant Treatment (Experimental): Following the completion of Arm 1, blood samples, flow-mediated dilation, lung function, and exercise capacity (VO2 peak) will be performed, only in patients with CF, at baseline, 4 weeks, 8 weeks, and 12 weeks following one of the following: 1) an anti-oxidant cocktail (vitamin C 1000 mg, vitamin E 400 IU, and alpha lipoic acid 600 mg) taken once a day, 2) 1500 mg Resveratrol once a day or 3) 10 mg Mitoquinol once a day.
  Interventions: Dietary Supplement: Chronic Antioxidant

INTERVENTIONS:
Dietary Supplement: Acute Antioxidant — Flow-Mediated Dilation will be determined at baseline and 2 hours following acute antioxidant treatment
  Other Names: Vitamin C; Vitamin E; Alpha Lipoic Acid; Resveratrol; Mitoquinol (MitoQ)
  Arms: Acute Antioxidant Treatment
Dietary Supplement: Chronic Antioxidant — Flow-Mediated Dilation will be determined at baseline, week 4, week 8, and week 12.
  Other Names: Vitamin C; Vitamin E; Alpha Lipoic Acid; Resveratrol; Mitoquinol (MitoQ)
  Arms: Chronic Antioxidant Treatment
Other: Placebo — Flow-Mediated Dilation will be determined at baseline and 2 hours following acute antioxidant treatment
  Arms: Acute Antioxidant Treatment

SUMMARY:
Cystic fibrosis has many health consequences. A reduction in the ability to perform exercise in patients with CF is related to greater death rates, steeper decline in lung function, and more frequent lung infections. However, the physiological mechanisms for this reduced exercise capacity are unknown. The investigators recently published the first evidence of systemic vascular dysfunction in patients with CF. Therefore, it is reasonable to suspect that the blood vessels are involved with exercise intolerance in CF. This study will look at how and if oxidative stress contributes to both artery dysfunction and exercise intolerance in CF.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is the most common fatal genetic disease in North America. The most disturbing aspect of CF is the associated premature death, most often due to respiratory complications. Clinical manifestations of CF include not only lung dysfunction, but many other systemic consequences as well. Systemic oxidative stress and exercise intolerance are established phenotypes in patients with CF. Additionally, for the first time the investigators have recently published the presence of systemic endothelial dysfunction in a cohort of young patients with CF who exhibited normal oxygen saturation and spirometric function.

Exercise intolerance, the limitation of the ability to perform exercise at the expected level, has been shown to predict mortality in patients with CF independent of lung function. Exercise capacity (VO2 peak), an objective measurement of exercise tolerance, drops approximately 5-8% per year in patients with CF. This excessive decay in exercise capacity not only leads to more pulmonary infections and deterioration of lung function, it represents a 5-8 fold decline compared to healthy sedentary adults. Preventing the excessive annual reduction in exercise capacity is essential to increasing the quality of life and longevity of patients with CF. However, a critical barrier to improving exercise capacity in CF is the investigators lack of knowledge regarding the different physiological mechanisms that contribute to exercise intolerance. It is important to emphasize that decreases in lung function (FEV1) do not always contribute to reductions in VO2 peak. Furthermore, less than 2% of patients who have an FEV1 greater than 50% predicted will have a significant drop in hemoglobin oxygen saturation (SpO2) during maximal exercise. These data suggest that mechanisms other than lung function induced hypoxemia may be contributing to exercise intolerance in patients with CF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF and healthy controls
* Men and women (> 18 yrs. old)
* Boys and girls (7-17 yrs. old)
* FEV1 percent predicted > 30%
* Patients with or without CF related diabetes
* Resting oxygen saturation (room air) >90%
* Traditional CF-treatment medications
* Ability to perform reliable/reproducible PFTs
* Clinically stable for 2 weeks (no exacerbations or need for antibiotic treatment within 2 weeks of testing or major change in medical status)
* Pancreatic sufficient and pancreatic insufficient patients

Exclusion Criteria:

* Children 6 yrs. old and younger
* FEV1 percent predicted < 30%
* Resting oxygen saturation (room air) < 90%
* Clinical diagnosis of heart disease, PAH
* Febrile illness within two weeks of visit
* Currently smoking, pregnant, or nursing
* Individuals on vaso-active medications (i.e. nitrates, beta blockers, ACE inhibitors, etc.)
* Patients with B. cepacia (only ~3% of our CF center patient population)
* Treatment for pulmonary exacerbation within 4 weeks of a study visit

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Acute Change in Flow mediated dilation | Change from baseline (2 hours)
  Flow-Mediated Dilation will be determined at baseline and 2 hours following acute antioxidant treatment
Chronic Change in Flow mediated dilation | Baseline, week 4, week 8, and week 12
  Flow-Mediated Dilation will be determined at baseline, week 4, week 8 and week 12.
Acute Change in exercise capacity (VO2 peak) | Baseline and 2 hours following acute antioxidant treatment
  Subjects will perform a baseline maximal exercise capacity test and on a separate visit perform a maximal exercise capacity test 2 hours following acute antioxidant treatment
Chronic Change in exercise capacity (VO2 peak) | Baseline, week 4, week 8, and week 12
  Subjects will perform a maximal exercise capacity test at baseline, week 4, week 8, and week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Harris, Ph.D., Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes